CLINICAL TRIAL: NCT06921629
Title: The Prevalence and Impact of Menstrual Complaints in Adolescents and Adults - a Prospective Cohort
Brief Title: Menstrual Complaints in Adolescents and Adults
Acronym: MEK app
Status: Active, not recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Dr. Robert A. de Leeuw, MD, PhD. Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: MEK-app
Record Dates: First submitted 2025-03-26; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Dysmenorrhea; Heavy Menstrual Bleeding; Daily Activities; Menstrual Cramps; Menstrual Cycle; Menstrual Distress (Dysmenorrhea); Menstrual Health Intervention; Menstrual Pain; Mobile Health; Mobile Health Technology (mHealth)
Keywords: Dysmenorrhea; Heavy Menstrual Bleeding; Menstrual complaints; Impact of menstrual complaints; daily activities; Adolescents; Adults
MeSH Terms: conditions — Dysmenorrhea; Menorrhagia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adolescents: postmenarchal adolescents between 12 and 18 years old, (according to the WHO's definition of adolescents) with monthly menstruation
  Interventions: Other: Menstruatie Educatie Kalender (Menstrution Education Calendar) application (MEK-app); Other: Questionnaires
- Adults: Postmenarchal adults between 19 and 60 years with monthly menstruation
  Interventions: Other: Menstruatie Educatie Kalender (Menstrution Education Calendar) application (MEK-app); Other: Questionnaires

INTERVENTIONS:
Other: Menstruatie Educatie Kalender (Menstrution Education Calendar) application (MEK-app) — The MEK-APP is a mHealth application to evaluate menstrual complaints like heavy menstrual blood loss and dysmenorrhea. The MEK-APP is a calendar and facilitates daily monitoring of pain intensity using a Visual Analogue Scale (VAS), the amount of blood loss through a pictorial blood loss assessment chart (PBAC), and the impact of these complaints on daily life. The MEK-APP followed the waterfall methodology for software development and the usability was evaluated by both adults and adolescents(4). Furthermore, the MEK app has been approved by the privacy and security officers of Amsterdam UMC
Other: Questionnaires — After registration for this study via www.mijnmenstruatie.nl (which has also been approved by the privacy and security officers of Amsterdam UMC), participants received the first digital questionnaire. This questionnaire consisted of a baseline questionnaire, the electronic self bleeding assessment tool (e-self-BATH) and the Menstrual Health Literacy questionnaire.
  After using the MEK-app for at least one month, participants received an e-mail with the second questionnaire. This questionnaire consisted of the Menstrual Bleeding Questionnaire; Period ImPact and Pain Assesment; Pelvic Pain Impact Questionnaire; ENDOPAIN-4D; Endometriosis Health Profile 5 and iMTA Productivity Cost Questionnaire.

SUMMARY:
The aim of this study is to investigate the prevalence of menstrual complaints and their impact on daily life activities (school/work absence, absence from social activities, sports) in adults and adolescents.

DETAILED DESCRIPTION:
This study was an online prospective cohort study and consisted of using the Menstruatie Educatie Kalender (Menstruation Education Calendar) application (MEK app) daily for at least one cycle with a questionnaire before and after the use of this application. Participants consisted of postmenarchal adolescents and adults with a menstrual cycle with monthly bleeding. The study involved minimal effort for participants: a baseline questionnaire at the start of the study, requiring approximately 10 minutes; daily app use for at least one cycle, taking around 20 seconds each day; and a final questionnaire at the end of the study, lasting about 10 minutes. Participants received no compensation for participating and the use of the MEK app was free.

Previous research on menstrual complaints in adolescents has considered sample sizes of approximately 1,000 participants to be representative of the population. Since this prospective cohort study about adolescent's menstrual complaints involved repeated measurements, and the literature suggested that repeated measurements of outcome variables increase study power and reduce the required sample size, this study aimed to include a total of 900 adolescents and 900 adults.

The study results were reported using descriptive statistical analyses. To compare dichotomous outcomes the chi-square test or the Fishers' exact test was used. Depending on the data distribution, the Student's t-test or Mann-Whitney U test was used to compare continuous outcomes. Mixed effects logistic regression was used for the association between menstrual complaints and the impact on daily life activities. The statistical analysis was performed in IBM SPSS Statistics version 28 using a two-sided p-values. P-values under 0.05 were considered statistically significant.

ELIGIBILITY:
The inclusion criteria were

* post-menarcheal adolescents and adults aged 12-60 years,
* having a menstrual cycle with monthly bleeding (also with an intra-uterine device or use of contraceptive pills),
* speaking Dutch (MEK-app is available in Dutch only);
* having a smartphone with the operating system Android or iOS and
* obtaining informed consent from the participant and the parents of the participants aged 12-16 years.

The exclusion criteria were

* amenorrhea
* incompleted questionnaires
* not using the MEK-app for at least one period

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants were recruited from social media channels Facebook (@Uterine Repair Center), Instagram (@MenstruatieApp) and Tiktok (@MenstruatieEducatieApp), schools during biology class and from outpatient clinics, including pediatrics and adolescent medicine and gynecology, regardless of their reason for coming.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2026-05-11 (Estimated); Study Completion 2026-05-11 (Estimated)

PRIMARY OUTCOMES:
Impact of menstrual complaints (registred in the MEK-app) | 1 month
  The impact of menstrual complaints (bleeding and pain) on daily activities in adolescents and adults registered in the MEK-app. Impact on daily life was assessed in the MEK app with the question: "Has your menstruation affected your daily activities?" Participants could respond with "yes" or "no."
Prevalence of menstrual complaints | 1 month
  Prevalence of dysmenorrhea and heavy menstrual bleeding

SECONDARY OUTCOMES:
Risk of clotting disorder (self-BAT questionnaire) | 1 month
  The risk of a clotting disorder, specifically in the groups with normal and heavy blood loss assessed with the self-BAT questionnaire. The results will be expressed as percentages of participants with increased self-BAT scores.
Knowledge about menstruation and management, measured with the Menstrual Health Literacy survey. | 1 month
  The Menstrual Health Literacy Survey consisted of questions about among other things current management options for dysmenorrhea, impact of dysmenorrhea and/or pelvic pain on daily or social activities, impact of dysmenorrhea on academic performance or engagement, school and/or university support, health literacy around menstruation, sources of knowledge, what they consider normal regarding dysmenorrhea, which additional symptoms during menstruation they perceive as normal, and how they manage the pain. The questionnaire was as a mixture of closed, multiple-choice, and open-ended questions. The answers to the questions in this questionnaire will be shown in numbers and percentages

CONTACTS AND LOCATIONS:
Overall Officials: Robert de Leeuw, MD, PhD, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ozcan H, Burger NB, Derksen ME, Peute LW, Huirne JAF, De Leeuw RA. The differences between adults and adolescents using a mobile health application for menstrual complaints: A usability and qualitative study. Int J Med Inform. 2024 May;185:105382. doi: 10.1016/j.ijmedinf.2024.105382. Epub 2024 Feb 23. PMID 38437753